CLINICAL TRIAL: NCT02032108
Title: Effects of Lifestyle Education Programs on Diabetes Control Among Diabetic Patients at Kigali University Teaching Hospital Rwanda
Brief Title: Effects of Lifestyle Education Programs on Diabetes Control in Rwanda
Acronym: LIDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kigali University Teaching Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Etienne Amendezo, Dr, Kigali University Teaching Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LID
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes lifestyle intervention Rwanda
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle counselling (Experimental): A 45-min lifestyle educational session will be delivered to the subjects randomized to the intervention group every month for one year.
  Lifestyle intervention will consist in group counselling on dietary habits, effects of regular physical activity, importance of adherence to medications, diabetes complications, actions to control blood sugar and ways of coping with stress.
  Interventions: Behavioral: lifestyle counselling

INTERVENTIONS:
Behavioral: lifestyle counselling — A 45-min lifestyle educational session will be delivered to the subjects randomized to the intervention group every month for one year.
  Lifestyle intervention will consist in group counselling on dietary habits, effects of regular physical activity, importance of adherence to medications, diabetes complications, actions to control blood sugar and ways of coping with stress.

SUMMARY:
Strategies to reduce the burden of diabetes in Rwanda, like in other resource poor settings, include involving diabetic patients in their own care and targeting modifiable risk factors through adopting appropriate dietary and lifestyle habits. According to previous research carried out in developed countries, lifestyle modifications may have effect on the development of diabetes and prevention of its complications.

However, direct evidence to show whether lifestyle intervention is beneficial for diabetic patients in resources limited countries like Rwanda is an open question. Though in these countries, access to healthy diet is claimed to be the barrier of implementation of therapeutic lifestyle based initiatives, we hypothesize that knowledge gaps are more important barriers than access to healthier diets and other lifestyle habits. We therefore would like to carry out this intervention to assess the effects of lifestyle education programs on glycemic control among people with diabetes followed up at CHUK.

DETAILED DESCRIPTION:
The study is a randomized controlled trial with two groups (one interventional and one control) to be followed up for 12 months. It will be carried out in Kigali University Teaching Hospital, the main referral hospital in Rwanda.

Lifestyle intervention will consist in group counselling on dietary habits (meals composition, importance and ways to reduce unhealthy foods: salty (especially because hypertension is of concern among diabetic people and blood pressure will be one of the secondary outcome measures), sugar, unsaturated fats, smoking, alcohol abuse and adapt healthier regimens including fruits & vegetables), effects of regular physical activity, importance of adherence to medications (including taking medications as directed, regular medical follow up,etc…), diabetes complications, actions to control blood sugar and ways of coping with stress.

Education & counselling sessions will be provided by a team of registered dietitians, nurses and counselors who will have been trained for this purpose prior to the intervention and will be taking between 45 to 60 min.

After baseline data collection, subjects in the control group will continue to receive usual care delivered by attending physicians and nutritionists at CHUK. This includes usual monthly medical follow up and individual conselling on dietary habits and lifestyle change delivered by attending physicians and/or dietitians

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes known since three months at least,
* being currently on treatment (insulin or oral hypoglycemiants),
* able to follow up at CHUK

Exclusion Criteria:

* patients with advanced diabetic complications (advanced nephropathy & CKD, proliferative retinopathy, recent history of myocardial infarction & severe Heart Failure (LVEF<35%), peripheral artery disease, stroke, severe diabetic foot disease,
* any other severe illness that may impede the patient's functional capacity,
* severe psychiatric disorders
* pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
between groups difference in glycated haemoglobin (HbA1c) | 12 months
  At the end of 12 months follow up, the mean (or median) differences in glycated hemoglobin of the interventional group and the control group will be analysed.

SECONDARY OUTCOMES:
endpoint versus baseline differences in glycated hemoglobin | 12 months
  at the end of 12 months follow up, endpoint versus baseline differences in the overall study population glycated hemoglobin levels will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte M. Bavuma, Dr, Study Chair — Kigali University Teaching Hospital; Etienne Amendezo, Dr, Principal Investigator — Kigali University Teaching Hospital
Locations (1):
- Kigali University Teaching Hospital, Kigali, Kigali, Rwanda

REFERENCES:
- [Derived] Amendezo E, Walker Timothy D, Karamuka V, Robinson B, Kavabushi P, Ntirenganya C, Uwiragiye J, Mukantagwabira D, Bisimwa J, Uwintwali Marie H, Umulisa H, Niyomwungeri S, Ndayambaje B, Dusabejambo V, Bavuma C. Effects of a lifestyle education program on glycemic control among patients with diabetes at Kigali University Hospital, Rwanda: A randomized controlled trial. Diabetes Res Clin Pract. 2017 Apr;126:129-137. doi: 10.1016/j.diabres.2017.02.001. Epub 2017 Feb 10. PMID 28237859